CLINICAL TRIAL: NCT00258882
Title: Post-licensure Safety Surveillance Study of Routine Use of Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (Adacel®)
Brief Title: Descriptive, Post-marketing, Passive Surveillance Safety Study of ADACEL™ Vaccine
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: TD512
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Pertussis
Keywords: Tetanus Toxoid,; acellular pertussis,; diphtheria toxoid
MeSH Terms: conditions — Whooping Cough; Tetanus | interventions — Tetanus Toxoid; Diphtheria Toxoid; adacel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Tetanus Toxoid, acellular pertussis, diphtheria toxoid — 0.5 mL, Intramuscular
  Other Names: Adacel®

SUMMARY:
To further characterize the vaccine safety profile and to identify any signals of potentially vaccine-related adverse events (AEs) not detected during pre-licensure studies.

DETAILED DESCRIPTION:
Surveillance using a healthcare organization with large comprehensive medical encounter databases will be used in this study to identify any risks or uncommon events associated with use of the recently licensed Adacel vaccine that may occur in routine clinical usage in a large population.

No investigational vaccines will be administered in this study. Participants will be included in the study on the basis of their having received Adacel vaccine as part of routine care.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of ADACEL vaccine during the study period

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Passive surveillance by review of Kaiser Permanente Medical Care Program (KPMCP) computerized records and state mortality tapes
Sampling Method: Probability Sample
Enrollment: 327293 (Actual)
Dates: Start 2006-01; Primary Completion 2011-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (3):
- United States (3):
  - Oakland, California
  - Aurora, Colorado
  - Portland, Oregon

REFERENCES:
- [Result] Baxter R, Hansen J, Timbol J, Pool V, Greenberg DP, Johnson DR, Decker MD. Post-licensure safety surveillance study of routine use of tetanus toxoid, reduced diphtheria toxoid and 5-component acellular pertussis vaccine. Hum Vaccin Immunother. 2016 Nov;12(11):2742-2748. doi: 10.1080/21645515.2016.1201622. Epub 2016 Jul 7. PMID 27388557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participant accrual occurred from 02 September 2005 through 16 October 2006 using 3 Kaiser Permanente databases.
Pre-assignment Details: Databases were reviewed to identify persons who received Adacel vaccine and Td vaccinated historical controls. Two statistical analysis methods were used, risk interval and historic cohort method. Adacel-exposed pregnancy cases were matched to non-exposed pregnant controls (3:1 ratio).
Groups:
- Adacel Vaccine Group: Participants who received Adacel vaccine during the study period were sub-grouped as 1) pregnant at the time of vaccination or who became pregnant within 28 days after vaccination and 2) non-pregnant recipients classified by age at vaccination.
- Control Groups: For each pregnant individual receiving Adacel vaccine, 3 control individuals not given Adacel vaccine were matched on age and month of their first positive pregnancy test. For non-pregnant individuals, age-matched individuals were identified who received Td vaccine but no live virus vaccine during the year prior to initiation of the study during the same month as Adacel vaccine recipient, but 1 year earlier.
Period: Adacel Recipients Historic Cohort Method
Arm/Group | Adacel Vaccine Group | Control Groups
Started | 124139 | 203154
Completed | 124139 | 203154
Not Completed | 0 | 0
Period: Adacel Recipients-Risk Interval Method
Arm/Group | Adacel Vaccine Group | Control Groups
Started | 124139 | 0 (Study participants served as their own controls for this analysis)
Completed | 124139 | 0
Not Completed | 0 | 0
Period: Pregnancy Surveillance
Arm/Group | Adacel Vaccine Group | Control Groups
Started | 225 (Adacel recipients who were pregnant at the time of vaccination or within 28 days thereafter.) | 675 (Non-vaccinated age-matched subjects with first positive pregnancy test in the same month (± 1 month))
Completed | 225 | 675
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received Adacel vaccine during the study period and age matched participants who received Td vaccine but no live virus vaccine, during the year prior to initiation of study during the same month as the Adacel vaccine recipient, 1 year earlier.
Groups:
- Adacel Vaccine Group: Participants who received Adacel vaccine during the study period were sub-grouped as 1) pregnant at the time of vaccination or who became pregnant within 28 days after vaccination and 2) non-pregnant recipients classified by age at vaccination.
  Each non-pregnant recipient served as their own control for evaluation of acute events. Rates of events occurring during Day 0 to 60 following vaccination were compared to rates of events occurring during Day 61 to 120 following vaccination (Short-term surveillance)
- Control Groups: Non-pregnant individuals matched by age to individuals who received Td vaccine but no live virus vaccine during the year prior to initiation of the study during the same month as Adacel vaccine recipient, but 1 year earlier.
- Total: Total of all reporting groups
Arm/Group | Adacel Vaccine Group | Control Groups | Total
Number analyzed (Participants) | 124139 | 203154 | 327293
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50214 | 58823 | 109037
  Between 18 and 65 years | 70861 | 119390 | 190251
  >=65 years | 3064 | 24941 | 28005
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.1 (19.0) | 39.0 (21.6) | 36.4 (20.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67067 | 104898 | 171965
  Male | 57072 | 98256 | 155328
Region of Enrollment [Number; unit: participants]
  United States | 124139 | 203154 | 327293
Seasonality (Time of vaccination) [Number; unit: Participants]
  December to February | 20293 | 42397 | 62690
  March to May | 35651 | 51039 | 86690
  June to August | 49173 | 62906 | 112079
  September to November | 19022 | 46812 | 65834

OUTCOME MEASURES:

1. Primary Outcome: Twenty One Pre-specified Outcomes of Interest as Obtained From International Coding of Diseases (ICD-9) Codes Captured After Adacel Vaccination in Clinical Database
Description: The twenty one pre-specified outcomes of special interest screened for in this study included: Arthritis, Arthralgia, or Arthropathy; Bell's Palsy; Diabetes; Encephalitis; Encephalopathy; Febrile Illness; Guillain-Barré; Hemolytic Anemia; Hypersensitivity; Idiopathic Thrombocytopenic Purpura (ITP); Lupus; Mixed Connective Tissue Disease; Multiple Sclerosis; Neuralgia; Neuritis; Neuropathy; Rheumatoid Arthritis; Scleroderma; Seizure; Severe Local Reaction; Transverse Myelitis.
  Comparison of events rates was performed using the risk-interval cohort design. In this design, the combined experience of individuals receiving Adacel vaccine served as their own control for evaluation of pre-specified outcomes of interest. Rates of events occurring during Days 0 to X (where X = 7, 14, 30, and 60) following vaccination were compared to rates of events occurring in the same individuals during Days 61 to 120 following vaccination.
Time Frame: Days 0 to 60 and Day 61 to 120 following vaccination
Population: Individuals receiving Adacel vaccine served as their own control for evaluation of acute events.
Measure: Number; unit: Events Per 1000 Person-months
Groups:
- Adacel Vaccine Group: Participants who received Adacel vaccine during the study period.
- Control Groups: Age matched participants who received Td vaccine but no live virus vaccine, during the year prior to initiation of study during the same month as the Adacel vaccine recipient, 1 year earlier.
Arm/Group | Adacel Vaccine Group | Control Groups
Number analyzed (Participants) | 124139 | 0
Events Per 1000 Person-months | 0 |

2. Primary Outcome: Twenty One Pre-specified Outcomes of Interest (ICD-9 Codes) Captured After Adacel Vaccination in Clinic Database
Description: The twenty one pre-specified outcomes of special interest screened for in this study included: Arthritis, Arthralgia, or Arthropathy; Bell's Palsy; Diabetes; Encephalitis; Encephalopathy; Febrile Illness; Guillain-Barré; Hemolytic Anemia; Hypersensitivity; ITP; Lupus; Mixed Connective Tissue Disease; Multiple Sclerosis; Neuralgia; Neuritis; Neuropathy; Rheumatoid Arthritis; Scleroderma; Seizure; Severe Local Reaction; Transverse Myelitis.
  Comparison of events rates was performed using the historic cohort design in which screening for possible new-onset chronic illnesses during the first 6 months following vaccination was performed. For each age-subgroup event, rates during the 6 months following vaccination among persons receiving Adacel vaccine were compared to event rates during the 6 months following vaccination among persons in the same age subgroup who received Td vaccine, but no live virus vaccine, during the year prior to initiation of this study.
Time Frame: Days 0 up to 180 following vaccination
Population: Individuals receiving Adacel vaccine served as their own control for evaluation of acute events.
Measure: Number; unit: Events Per 1000 Person-months
Arm/Group | Adacel Vaccine Group | Control Groups
Number analyzed (Participants) | 124139 | 203154
Events Per 1000 Person-months | 0 | 0

3. Primary Outcome: All Diagnoses (Coded as ICD-9 Codes) Occurring During Specific Periods After Vaccination in All Adacel Exposed Individuals in Emergency Department and Hospital Databases.
Description: Surveillance for acute onset outcomes occurring shortly (days to weeks) after vaccination was performed using the risk-interval cohort design. In this design, the combined experience of individuals receiving Adacel vaccine served as their own control for evaluation of acute events. Rates of events occurring during Days 0 to X (where X = 7, 14, 30, and 60) following vaccination were compared to rates of events occurring in the same individuals during Days 61 to 120 following vaccination
Time Frame: Days 0 to 60 and Day 61 to 120 following vaccination
Population: Individuals receiving Adacel vaccine served as their own control for evaluation of acute events.
Measure: Number; unit: Events Per 1000 Person-months
Arm/Group | Adacel Vaccine Group | Control Groups
Number analyzed (Participants) | 124139 | 0
Events Per 1000 Person-months | 0 |

4. Primary Outcome: All Diagnoses (Coded as ICD-9 Codes) Occurring During 6 Months After Vaccination in All Adacel Exposed Individuals in Emergency Department and Hospital Databases.
Description: Comparison of events rates was performed using the historic cohort design in which screening for possible new-onset chronic illnesses during the first 6 months following vaccination was performed. For each age-subgroup event, rates during the 6 months following vaccination among persons receiving Adacel vaccine were compared to event rates during the 6 months following vaccination among persons in the same age subgroup who received Td vaccine, but no live virus vaccine, during the year prior to initiation of this study.
Time Frame: Days 0 to 180 following vaccination
Population: Individuals receiving Adacel vaccine served as their own control for evaluation of acute events.
Measure: Number; unit: Events per 1000 Person-months
Arm/Group | Adacel Vaccine Group | Control Groups
Number analyzed (Participants) | 124139 | 0
Events per 1000 Person-months | 0 |

5. Primary Outcome: Summary of Maternal Outcomes in Pregnant Adacel Recipients and Pregnant Non-Adacel Recipient Controls
Description: Pregnancies were identified by positive pregnancy tests or prenatal visits within 9 months prior to vaccination with no record of pre-vaccination delivery or abortion, or by prenatal visits, therapeutic abortions, or deliveries within 10 months after vaccination. For all such pregnancies, further review (including chart review, provider and vaccinee interviews, or other appropriate steps) was conducted to identify those for whom it could not be excluded that the individual was pregnant at the time of vaccination or within 28 days thereafter. Such pregnancies were reported by Kaiser Permanente Vaccine Study Center to the Adacel Pregnancy Registry. Maternal and fetal outcomes (up to 1 month of life) were enumerated. For each pregnant Adacel vaccine subjects, 3 age-matched non-Adacel vaccinated controls (± 1 year) that had a first positive pregnancy test during the same month (± 1 month). Rates of events of maternal and fetal outcomes were compared between the 2 groups.
Time Frame: Pregnancy to Delivery, up to 9 months
Population: All persons in the database searches as being vaccinated with Adacel vaccine during pregnancy or within 28 days prior to becoming pregnant and age-matched pregnant controls who did not receive Adacel vaccine.
Measure: Number; unit: Participants
Groups:
- Adacel Vaccine Group: Participants who received Adacel vaccine during the study period and were pregnant at the time of vaccination or became pregnant within 28 days after vaccination.
- Control Groups: Age matched pregnant controls who did not receive Adacel vaccine.
Arm/Group | Adacel Vaccine Group | Control Groups
Number analyzed (Participants) | 225 | 675
Participants
  Life Birth | 165 | 442
  Spontaneous abortion (<20 weeks gestation) | 21 | 102
  Early fetal death (20-27 weeks gestation) | 0 | 1
  Late fetal death (at least 28 weeks gestation) | 1 | 0
  Elective abortion | 33 | 105
  Ectopic pregnancy | 1 | 5
  Lost to follow-up | 4 | 20

6. Primary Outcome: Summary of Fetal Outcomes in Infants Born to Adacel Exposed Pregnant Women and Infants Born to Non-Adacel Exposed Pregnant Controls.
Description: as for outcome 5
Time Frame: Pregnancy to Delivery, up to 9 months
Population: as for outcome 5
Measure: Number; unit: Infants
Arm/Group | Adacel Vaccine Group | Control Groups
Number analyzed (Participants) | 225 | 675
Infants
  Encephalocele | 1 | 0
  Specified congenital anomalies of lacrimal passage | 4 | 18
  Ventricular septal defect | 1 | 2
  Stenosis of pulmonary valve, congenital | 0 | 1
  Patent ductus arteriosus | 2 | 6
  Agenesis, hypoplasia, and dysplasia of lung | 0 | 1
  Cleft palate, unilateral, incomplete | 0 | 1
  Cleft palate with cleft lip, unspecified | 0 | 1
  Tongue tie | 1 | 6
  Undescended testis | 0 | 1
  Hypospadias | 2 | 0
  Congenital chordee | 0 | 2
  Other penile anomalies | 0 | 2
  Other obstructive defects of renal pelvis and uret | 1 | 0
  Metatarsus varus | 1 | 0
  Polydactyly of fingers | 0 | 1
  Polydactyly of toes | 0 | 1
  Other congenital deformity of hip (joint) | 0 | 1
  Vascular hamartomas | 1 | 2
  Congenital pigmentary anomalies of skin | 1 | 5
  Other specified anomalies of skin | 0 | 2
  Specified congenital anomalies of breast | 0 | 1
  Down's syndrome | 0 | 1
  Congenital anomaly, unspecified | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events data surveillance period were only in Adacel vaccine recipients from the day of vaccination up to 6 months post-vaccination from the Outpatient, Emergency Room and Hospital databases.
Description: Total number reported for the serious adverse events are events that were deemed possibly associated with the Adacel vaccine in the Outpatient, Emergency Room and Hospital databases.
Groups:
- Adacel Vaccine Group: Participants who received Adacel vaccine during the study period. They are sub-grouped as those pregnant at the time of vaccination with Adacel or who became pregnant within 28 days after vaccination and other recipients are classified by age at vaccination.
Arm/Group | Adacel Vaccine Group
Serious Adverse Events (participants affected / at risk) | 4/124139
Other Adverse Events (participants affected / at risk) | 0/124139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adacel Vaccine Group (N=124139)
Bell Palsy (Nervous system disorders) | 2
Guillain-Barré syndrome (Musculoskeletal and connective tissue disorders) | 1
Epilepsy (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
As a result of screening using The Risk Interval and The Historic Cohort methods incident rates for 1030 outcomes were flagged as elevated. In post-hoc manual review no safety signals were identified. Details highlighted in the manuscript.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.